CLINICAL TRIAL: NCT01280578
Title: The Coherex PFO Migraine Registry
Brief Title: The Coherex FlatStent™ EF PFO Migraine Registry
Status: Terminated | Type: Observational
Why Stopped: Lack of enrollment
Sponsor: Coherex Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: RESPONDER
Record Dates: First submitted 2011-01-19; First posted 2011-01-21 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Patients With Migraine and PFO
Keywords: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Transcatheter PFO Closure — Transcatheter PFO Closure
  Other Names: Coherex FlatStent™ EF PFO Closure System

SUMMARY:
A prospective, single arm, multicenter clinical registry evaluating the change in migraine headaches in migraine with aura patients who undergo patent foramen ovale (PFO) closure with the Coherex FlatStent™ EF PFO Closure System.

ELIGIBILITY:
Major Inclusion Criteria:

Age 18-65 males and non pregnant females History of refractory migraine Documented PFO

Major Exclusion Criteria:

Known allergy to aspirin or nickel. Medication Overuse Headache Body mass index > 40. Recent Botulinum neurotoxin type A treatment Other known structural heart disease, coronary artery disease, atrial fibrillation PFO morphology not suitable for FlatStent EF Patients who have had a stroke within the past two months Post-traumatic headache. Patients with diagnosed hypercoagulable states that require chronic treatment with warfarin.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NA. Study terminated
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2011-02-01 (Actual); Primary Completion 2012-06-01 (Actual); Study Completion 2012-06-01 (Actual)

PRIMARY OUTCOMES:
Efficacy
  Percentage of subjects treated with the FlatStent EF who, achieve a clinically significant reduction in migraine or probable migraine headache days at follow-up.

SECONDARY OUTCOMES:
Closure efficacy
  Degree of closure of PFO at follow-up